CLINICAL TRIAL: NCT01125345
Title: A Prospective Controlled Clinical Trial to Evaluate the Posterior Capsule Opacification in Contralateral Eyes Implanted With Single Piece Hydrophobic AcrySof IOL and Single Piece Hydrophilic Acrylic IOLs
Brief Title: Posterior Capsule Opacification (PCO) With Single Piece Hydrophobic Versus Hydrophillic Intraocular Lens (IOL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Dr. Shetal M. Raj, Raghudeep Eye Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06-009
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-05

CONDITIONS: Posterior Capsule Opacification
Keywords: hydrophobic acrylic; PCO; posterior capsule opacification; hydrophilic acrylic IO
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hydrophobic IOL (Experimental): The single piece Acrysof hydrophobic IOL model- SN60WF
  Interventions: Procedure: Phacoemulsification
- Hydrophilic IOL (Active Comparator): Rayner Intraocular Lenses Ltd., England, Model C-flex 570C
  Interventions: Procedure: Phacoemulsification
- Hydrophillic IOL (Active Comparator): Bausch and Lomb ltd, model Akreos Adapt
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — Phacoemulsification with IOL implantation in eyes undergoing bilateral cataract surgery

SUMMARY:
The purpose of the study was to compare the postoperative PCO results of the single-piece hydrophobic Acrylic IOLs versus the newer generation single-piece hydrophilic Acrylic IOLs in patients undergoing bilateral cataract surgery.

DETAILED DESCRIPTION:
Amongst several surgical techniques and IOL technology that influence the opacification of the posterior capsule, the role of IOL material and optic design remain crucial in determining its development. The single-piece Acrylic IOLs with a hydrophobic surface have been widely used in practice. The single-piece Acrylic IOLs with a hydrophilic surface became commercially available more recently. Although there is a study that compared the single piece hydrophobic and the single piece hydrophilic IOL, it was conducted on the older generation of the hydrophilic IOL. Moreover, experimental and clinical study has been performed to evaluate the posterior capsule opacification between the Hydrophilic acrylic IOL with a sharp optic edge design excluding the optic-haptic junction, versus the newer generation hydrophilic IOL design which has an improved 360-degree sharp edge, with results favouring the latter design. There is little data that compares the single-piece Acrylic IOLs with a hydrophobic surface to the newer generation single-piece Acrylic IOLs with a hydrophilic surface. Because the IOL characteristics play a crucial role to prevent posterior capsule opacification (PCO), it is of clinical importance, as well as investigational interest to assess the PCO following implantation of these IOLs. We conducted a prospective, randomised, intra-individual study to compare the 3 year postoperative PCO results of the single-piece hydrophobic Acrylic IOLs versus the newer generation single-piece hydrophilic Acrylic IOLs in patients undergoing bilateral cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* bilateral senile surgery
* age ranged from 53 to 78 years
* pupil mydriasis > 7 mm
* No history of previous ocular surgery
* gave consent for followup examination

Exclusion Criteria:

* coexisting ocular morbidities
* diabetes mellitus

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
posterior capsule evaluation | 3 years

SECONDARY OUTCOMES:
ND-Yag capsulotomy rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Vasavada, MD, Principal Investigator — Iladevi Cataract and IOL Research Center
Locations (1):
- Raghudeep Eye Clinic, Ahmedabad, Gujarat, India

REFERENCES:
- [Background] Johansson B. Clinical consequences of acrylic intraocular lens material and design: Nd:YAG-laser capsulotomy rates in 3 x 300 eyes 5 years after phacoemulsification. Br J Ophthalmol. 2010 Apr;94(4):450-5. doi: 10.1136/bjo.2009.166181. Epub 2009 Oct 14. PMID 19828518
- [Background] Lombardo M, Carbone G, Lombardo G, De Santo MP, Barberi R. Analysis of intraocular lens surface adhesiveness by atomic force microscopy. J Cataract Refract Surg. 2009 Jul;35(7):1266-72. doi: 10.1016/j.jcrs.2009.02.029. PMID 19545819
- [Background] Kugelberg M, Wejde G, Jayaram H, Zetterstrom C. Two-year follow-up of posterior capsule opacification after implantation of a hydrophilic or hydrophobic acrylic intraocular lens. Acta Ophthalmol. 2008 Aug;86(5):533-6. doi: 10.1111/j.1600-0420.2007.01094.x. Epub 2007 Dec 11. PMID 18081899
- [Background] Kugelberg M, Wejde G, Jayaram H, Zetterstrom C. Posterior capsule opacification after implantation of a hydrophilic or a hydrophobic acrylic intraocular lens: one-year follow-up. J Cataract Refract Surg. 2006 Oct;32(10):1627-31. doi: 10.1016/j.jcrs.2006.05.011. PMID 17010858
- [Background] Heatley CJ, Spalton DJ, Kumar A, Jose R, Boyce J, Bender LE. Comparison of posterior capsule opacification rates between hydrophilic and hydrophobic single-piece acrylic intraocular lenses. J Cataract Refract Surg. 2005 Apr;31(4):718-24. doi: 10.1016/j.jcrs.2004.08.060. PMID 15899448
- [Background] Werner L, Mamalis N, Pandey SK, Izak AM, Nilson CD, Davis BL, Weight C, Apple DJ. Posterior capsule opacification in rabbit eyes implanted with hydrophilic acrylic intraocular lenses with enhanced square edge. J Cataract Refract Surg. 2004 Nov;30(11):2403-9. doi: 10.1016/j.jcrs.2004.02.085. PMID 15519096
- [Background] Nishi Y, Rabsilber TM, Limberger IJ, Reuland AJ, Auffarth GU. Influence of 360-degree enhanced optic edge design of a hydrophilic acrylic intraocular lens on posterior capsule opacification. J Cataract Refract Surg. 2007 Feb;33(2):227-31. doi: 10.1016/j.jcrs.2006.10.020. PMID 17276262